CLINICAL TRIAL: NCT00983242
Title: A One-Directional, Open Label Drug Interaction Study to Investigate the Effects of Multiple Dose Verapamil HCl ER on Single Dose Pharmacokinetics of Colchicine in Healthy Volunteers
Brief Title: Drug-Drug Interaction Between Colchicine and Verapamil ER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-08-1014
Record Dates: First submitted 2009-08-13; First posted 2009-09-24 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2009-10-15 (Estimated); Status verified 2009-10

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Colchicine; Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine alone (Active Comparator): baseline colchicine pharmacokinetics
  Interventions: Drug: Colchicine
- Colchicine with Verapamil HCl ER (Experimental): colchicine pharmacokinetics in presence of steady-state verapamil
  Interventions: Drug: Verapamil HCl ER; Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — A single dose of 0.6 mg colchicine administered alone at 8am on Day 1 after an overnight fast of at least 10 hours.
  Arms: Colchicine alone
Drug: Verapamil HCl ER — One 240 mg verapamil HCl ER tablet taken at 8am on Days 15-18 without regard to meals and along with colchicine at 8am on Day 19 after an overnight fast of at least 10 hours.
  Arms: Colchicine with Verapamil HCl ER
Drug: Colchicine — A single dose of 0.6 mg colchicine administered along with verapamil HCL ER at 8 am on Day 19 after an overnight fast of at least 10 hours.
  Arms: Colchicine with Verapamil HCl ER

SUMMARY:
Colchicine is a substrate for both cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp). Verapamil hydrochloride is a potent inhibitor of cytochrome P450 (CYP) 3A4 and P-gp. This study will evaluate the effect of multiple doses of extended-release verapamil hydrochloride (verapamil HCl ER) on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period.

DETAILED DESCRIPTION:
Colchicine is a substrate for both cytochrome P450 3A4 (CYP3A4) and P-glycoprotein (P-gp). Verapamil hydrochloride is a potent inhibitor of cytochrome P450 (CYP) 3A4 and P-gp. This study will evaluate the effect of multiple doses of extended-release verapamil hydrochloride (verapamil HCl ER) on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. On study Day 1 after a fast of at least 10 hours, twenty-four healthy, non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given one dose of colchicine (1 x 0.6 mg tablet). Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for 24 hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of colchicine. Blood sampling will then continue on a non-confined basis on Days 2-5. After a 14 day washout period, on Day 15 subjects will return to the clinic for dosing of verapamil HCl ER (1 x 240 mg tablet) and a post-dose confinement period of 12 hours. Subjects will return on Days 16-19 for a morning dose of verapamil HCl ER (1 x 240 mg tablet). Verapamil HCl ER doses administered on Days 15-18 will not necessarily be in a fasted state. On the morning of Day 19 after a fast of at least 10 hours, all study participants will receive co-administered single doses of colchicine (1 x 0.6 mg) and verapamil HCl ER (1 x 240 mg). Fasting will continue for 4 hours following these doses and subjects will be confined to the clinic for dosing and for 24 hours after the dose. Blood samples will be drawn at times sufficient to adequately define the pharmacokinetics of colchicine in the presence of verapamil HCL at steady state. Blood sampling will continue on a non-confined basis on Days 20-23. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Vital signs (blood pressure and pulse) will be measured pre-dose and 1, 2, and 3 hours post-dose on Day 1, pre-dose and 12 hours post-dose on Day 15, and pre-dose and 1, 2 ,3 and 12 hours post-dose on Day 19 to coincide with peak plasma concentrations of both colchicine and verapamil HCl ER. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age, non-smoking and non-pregnant (post-menopausal, surgically sterile or using effective contraceptive measures) with a body mass index (BMI) greater than or equal to 18 and less than or equal to 32, inclusive.

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation or plasma donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gallbladder or biliary tract, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease
* Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study
* Drug allergies to colchicine or verapamil

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-09; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, PharmD, Principal Investigator — PRACS - Cetero
Locations (1):
- PRACS Institute, Ltd. - Cetero Research, East Grand Forks, Minnesota, United States

REFERENCES:
- [Derived] Terkeltaub RA, Furst DE, Digiacinto JL, Kook KA, Davis MW. Novel evidence-based colchicine dose-reduction algorithm to predict and prevent colchicine toxicity in the presence of cytochrome P450 3A4/P-glycoprotein inhibitors. Arthritis Rheum. 2011 Aug;63(8):2226-37. doi: 10.1002/art.30389. PMID 21480191
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four (24) healthy, non-smoking, adult male and female volunteers consisting of the community at large were enrolled.
Pre-assignment Details: Forty-four (44) subjects were screened, thirteen (13) were screen failures, five (5) were transferred to a different study, one (1) did not appear at check in at Period 1 and one (1) was not needed for the study.
Groups:
- Colchicine Alone, Colchicine With Verapamil HCl ER: All subjects received each of the study treatments. At 8am on Day 1 after a 10 hour fast all subjects received a single dose of colchicine 0.6 mg followed by a 14 day washout period. At 8am on Days 15-18 all subjects received a dose of verapamil hydrochloride extended-release (verapamil HCl ER) 240 mg without regard to meals. At 8am on Day 19 after a fast of at least 10 hours all subjects received a single dose of colchicine 0.6 mg along with the final dose of verapamil HCl ER 240 mg.
Period: Colchicine Alone
Arm/Group | Colchicine Alone, Colchicine With Verapamil HCl ER
Started | 24
Completed | 24
Not Completed | 0
Period: 14 Day Washout Period
Arm/Group | Colchicine Alone, Colchicine With Verapamil HCl ER
Started | 24
Completed | 24
Not Completed | 0
Period: Verapamil HCl ER Alone
Arm/Group | Colchicine Alone, Colchicine With Verapamil HCl ER
Started | 24
Completed | 24
Not Completed | 0
Period: Colchicine With Verapamil HCl ER
Arm/Group | Colchicine Alone, Colchicine With Verapamil HCl ER
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Colchicine Alone, Colchicine With Verapamil HCl ER
Number analyzed (Participants) | 24
Age, Customized [Number; unit: participants] — >=18 and <=45
  participants
    <=18 years | 2
    Between 18 and 65 years | 22
    >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.75 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: On Days 1 and 19 - serial pharmacokinetic blood samples were collected pre-dose and at 0.5, 1.0, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, and 96 hours post-dose.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Colchicine Alone: At 8am on Day 1 after a fast of at least 10 hours all subjects received a single dose of colchicine 0.6 mg followed by a 14 day washout period.
- Colchicine With Verapamil HCl ER: At 8am on Days 15-18 subjects were administered verapamil hydrochloride extended release (verapamil HCl ER) 240mg without regard to meals. At 8am on Day 19 after a fast of at least 10 hours all subjects received a single dose of colchicine 0.6 mg along with the final dose of verapamil HCl ER 240mg.
Arm/Group | Colchicine Alone | Colchicine With Verapamil HCl ER
Number analyzed (Participants) | 24 | 24
pg/mL | 2,968.42 (1,259.63) | 3,850.63 (1,458.96)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the plasma concentration versus time curve beginning from the first dose (time 0) to the last measurable colchicine concentration (time t), as calculated by the linear trapezoidal method.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Verapamil HCl ER
Number analyzed (Participants) | 24 | 24
pg-hr/mL | 13,085.26 (5,292.05) | 24,637.91 (6,556.67)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable colchicine plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Verapamil HCl ER
Number analyzed (Participants) | 24 | 24
pg-hr/mL | 15,371.17 (6,311.09) | 30,586.33 (8,283.83)

ADVERSE EVENTS:
Groups:
- Colchicine Alone: At 8am on Day 1 after a 10 hour fast all subjects received a single dose of colchicine 0.6 mg followed by a 14 day washout period.
- Verapamil HCl ER: At 8am on Days 15-18 all subjects received a dose of verapamil HCl ER 240 mg without regard to meals.
- Colchicine With Verapamil HCl ER: At 8am on Day 19 following a 10 hour fast all subjects received one dose of verapamil HCl ER 240 mg along with one dose of colchicine 0.6 mg.
Arm/Group | Colchicine Alone | Verapamil HCl ER | Colchicine With Verapamil HCl ER
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 5 | 9 | 5
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Colchicine Alone | Verapamil HCl ER | Colchicine With Verapamil HCl ER
Abdominal pain upper (Gastrointestinal disorders) | 1/24 (1) | 0/24 (0) | 0/24 (0)
Constipation (Gastrointestinal disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Diarrhea (Gastrointestinal disorders) | 1/24 (1) | 0/24 (0) | 0/24 (0)
Nausea (Gastrointestinal disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Feeling hot (General disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1/24 (1) | 0/24 (0) | 0/24 (0)
Dizziness (Nervous system disorders) | 1/24 (1) | 0/24 (0) | 1/24 (1)
Headache (Nervous system disorders) | 3/24 (3) | 8/24 (13) | 4/24 (5)
Sinus congestion (Nervous system disorders) | 0/24 (0) | 1/24 (1) | 0/24 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days